CLINICAL TRIAL: NCT00527176
Title: Pulse Corticosteroid Therapy and Effect on Brain Water Diffusivity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Other Study IDs: B40320072108
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Corticosteroid; Pulse therapy; Diffusion weighted imaging; q Space Imaging
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In daily clinical use, pulse high dosis corticosteroids are used to treat cerebral edema in different pathological situations ( surgery, trauma, tumors...). Dehydration can theorically concern extra-cellular or intracellular water, or both.

The relative proportion of those two components are not known, as well their kinetics.

Diffusion Weighted Imaging ( DWI) is a none invasive and none toxic technique to study those phenomena.We can also study the diffusivity anisotropy not using a Gaussian distribution but rather a non- gaussian one, more close to the reality ( q Space Imaging ).

Finally, we can study the compartment redistribution between slow and rapid water molecules diffusion by bi-exponential decomposition of the diffusion signal, corresponding, theorically, respectively to the intra- and extra-cellular component.

Hypothesis : The high dosis steroid pulse therapy modifies or not the water free diffusion in DWI and qSI ? Is there a modification in the diffusivity of both rapid and slow component ?

ELIGIBILITY:
Inclusion Criteria:

* Systemic Lupus Erythematosus
* normal neurological exam
* informed consent
* 18 yo or more

Exclusion Criteria:

* abnormal neurological exam
* younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-09; Study Completion 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Duprez, MD, Study Director — UNIVERSITE CATHOLIQUE DE LOUVAIN; Denis Rommel, MD, Principal Investigator — UNIVERSITE CATHOLIQUE DE LOUVAIN
Locations (1):
- Clinique Universitaire St LUC, Brussels, Belgium

REFERENCES:
- [Background] Bosma GP, Huizinga TW, Mooijaart SP, Van Buchem MA. Abnormal brain diffusivity in patients with neuropsychiatric systemic lupus erythematosus. AJNR Am J Neuroradiol. 2003 May;24(5):850-4. PMID 12748084
- [Background] Moritani T, Shrier DA, Numaguchi Y, Takahashi C, Yano T, Nakai K, Zhong J, Wang HZ, Shibata DK, Naselli SM. Diffusion-weighted echo-planar MR imaging of CNS involvement in systemic lupus erythematosus. Acad Radiol. 2001 Aug;8(8):741-53. doi: 10.1016/S1076-6332(03)80581-0. PMID 11508753
- [Background] Steens SC, Steup-Beekman GM, Bosma GP, Admiraal-Behloul F, Olofsen H, Doornbos J, Huizinga TW, van Buchem MA. The effect of corticosteroid medication on quantitative MR parameters of the brain. AJNR Am J Neuroradiol. 2005 Nov-Dec;26(10):2475-80. PMID 16286387
- [Background] Dehmeshki J, Van Buchem MA, Bosma GP, Huizinga TW, Tofts PS. Systemic lupus erythematosus: diagnostic application of magnetization transfer ratio histograms in patients with neuropsychiatric symptoms--initial results. Radiology. 2002 Mar;222(3):722-8. doi: 10.1148/radiol.2223010413. PMID 11867791
- [Background] Peterson PL, Howe FA, Clark CA, Axford JS. Quantitative magnetic resonance imaging in neuropsychiatric systemic lupus erythematosus. Lupus. 2003;12(12):897-902. doi: 10.1191/0961203303lu499oa. PMID 14714908
- [Background] Moritani T, Hiwatashi A, Shrier DA, Wang HZ, Numaguchi Y, Westesson PL. CNS vasculitis and vasculopathy: efficacy and usefulness of diffusion-weighted echoplanar MR imaging. Clin Imaging. 2004 Jul-Aug;28(4):261-70. doi: 10.1016/S0899-7071(03)00191-8. PMID 15246475
- [Background] Sun SS, Huang WS, Chen JJ, Chang CP, Kao CH, Wang JJ. Evaluation of the effects of methylprednisolone pulse therapy in patients with systemic lupus erythematosus with brain involvement by Tc-99m HMPAO brain SPECT. Eur Radiol. 2004 Jul;14(7):1311-5. doi: 10.1007/s00330-003-2166-3. Epub 2003 Dec 9. PMID 14663624